CLINICAL TRIAL: NCT01924442
Title: CSP #517-FS - ROOBY Trial Extension (Randomized on Pump and Off Pump Bypass Surgery: Long Term Follow-up)
Brief Title: ROOBY Trial Follow-up Extension
Status: Completed | Type: Observational
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: 517-FS
Record Dates: First submitted 2013-07-18; First posted 2013-08-16 (Estimated); Results first posted 2019-06-07 (Actual); Last update posted 2019-06-07 (Actual); Status verified 2019-03

CONDITIONS: All Cause Mortality; MACE
Keywords: Coronary Artery Disease; Off-Pump; Myocardial Ischemia; Heart Disease
MeSH Terms: conditions — Coronary Artery Disease; Myocardial Ischemia; Heart Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- On-Pump: Cardiac bypass using Heart Lung Machine
- Off-Pump: Cardiac bypass surgery on beating heart

SUMMARY:
The Department of Veterans Affairs "Randomized On/Off Bypass" (ROOBY) Trial (CSP #517) was funded in 2001. ROOBY was designed to compare the short-term (30-day) and intermediate-term (1-year) outcomes for patients undergoing off-pump versus on-pump coronary artery bypass graft (CABG) procedures. The ROOBY trial reported a significantly higher 1-year adverse composite outcome rate (i.e., all-cause death, non-fatal myocardial infarction (MI) and/or repeat revascularization) for off-pump versus on-pump patients. ROOBY documented that a higher percentage of off-pump patients received fewer grafts than originally planned (i.e., off-pump patients were less completely revascularized) as compared to on-pump patients. Across all anatomic regions of the heart, the 1-year graft patency rates were significantly lower for off-pump CABG patients. Based on these ROOBY trial initial findings, critically important clinical questions related to the long-term efficacy, stability and durability of the off-pump versus on-pump techniques have been raised. Extending the original ROOBY trial, this CSP #517 follow-up study (CSP 517-FS) will evaluate the longer-term impact of off-pump versus on-pump surgical approaches upon the future occurrence of major adverse cardiovascular events (MACE).

DETAILED DESCRIPTION:
A debate is ongoing as to the potential longer-term benefits of off-pump versus on-pump treatments. A recent meta-analysis summarized 12 randomized trials with follow-up extending beyond 1-year; with a significant increase documented in the late off-pump repeat revascularization and mortality rates. As a very large single center study with longer-term follow-up, a Beijing hospital study reported that their early minor advantages identified for off-pump surgery (n = 3,266) were offset at 4.5 years by an increased risk for cardiac death, acute MI and repeat revascularization as compared to an on-pump (n = 3,399) approach. The OCTOPUS study (a multi-center randomized trial based in the Netherlands) concluded that there was no difference in off-pump versus on-pump procedures for 5-year cardiac outcomes. However, OCTOPUS critics raised questions as to whether this study of only 281 low-risk patients was adequately powered to detect 5-year clinically relevant differences.

The ROOBY trial represents the only US-based, multi-center trial that will be adequately powered to detect clinically relevant, statistically significant differences in these long-term MACE (i.e., all cause mortality, non-fatal myocardial infarction, and/or repeat revascularization) outcomes. Recognized as a landmark study, ROOBY has resulted in important contributions including 10 manuscripts, 2 letters to the editor, and an invited editorial. As of October 11, 2012, over 182 manuscripts (not including any self-citations) had referenced the ROOBY trial's original 2009 publication. Most recently, the ROOBY trial was identified in the 2012 Almanac of adult cardiac surgery, where the national society journals present selected research that has driven recent clinical care advances. Additionally, ROOBY was judged independently by the March 2012 Cochrane systematic review as one of only three, multi-center trials that had been conducted to-date with a low risk of bias.

The original ROOBY trial's enrollment was initiated in February 2002 and ended in June 2007. Given the passage of time, it is now possible to obtain at least 5 years of follow-up to identify these critically important longer-term MACE endpoints for all ROOBY patients. For the earliest ROOBY patients enrolled, their MACE outcomes for up to (and potentially beyond) 10 years post-CABG may be assessed. These MACE endpoints will be ascertained using a combination of VA and non-VA database extracts as well as by chart reviews. In summary, the CSP 517-FS proposed study represents the first, large scale, US-based, multi-center, randomized, controlled off-pump versus on-pump trial that will have adequate power to assess major adverse cardiovascular events beyond 5 years - comparing the long-term effectiveness of these procedures to guide future adult cardiac surgical clinical decision-making processes.

The Department of Veterans Affairs "Randomized On/off Bypass" (ROOBY) Trial (CSP#517; NCT00032630) was funded in 2001.

ELIGIBILITY:
Inclusion Criteria:

* All patients that survived to 1 year enrolled in the ROOBY Trial

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: To be eligible for the ROOBY trial, subjects were elective or urgent Coronary Artery Bypass only procedure candidates
Sampling Method: Non-Probability Sample
Enrollment: 2203 (Actual)
Dates: Start 2013-10-01 (Actual); Primary Completion 2016-09-01 (Actual); Study Completion 2018-09-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Annie Laurie Shroyer, PhD MHSA, Study Chair — Northport VA Medical Center, Northport, NY
Locations (1):
- Northport VA Medical Center, Northport, NY, Northport, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Quin JA, Wagner TH, Hattler B, Carr BM, Collins J, Almassi GH, Grover FL, Shroyer AL. Ten-Year Outcomes of Off-Pump vs On-Pump Coronary Artery Bypass Grafting in the Department of Veterans Affairs: A Randomized Clinical Trial. JAMA Surg. 2022 Apr 1;157(4):303-310. doi: 10.1001/jamasurg.2021.7578. PMID 35171210
- [Derived] Shroyer AL, Hattler B, Wagner TH, Collins JF, Baltz JH, Quin JA, Almassi GH, Kozora E, Bakaeen F, Cleveland JC Jr, Bishawi M, Grover FL; Veterans Affairs ROOBY-FS Group. Five-Year Outcomes after On-Pump and Off-Pump Coronary-Artery Bypass. N Engl J Med. 2017 Aug 17;377(7):623-632. doi: 10.1056/NEJMoa1614341. PMID 28813218

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | On-Pump | Off-Pump
Started | 1099 | 1104
Completed | 1059 | 967
Not Completed | 40 | 137

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | On-Pump | Off-Pump | Total
Number analyzed (Participants) | 1099 | 1104 | 2203
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 699 | 671 | 1370
  >=65 years | 400 | 433 | 833
Age, Continuous [Mean (Standard Deviation); unit: Years] | 62.5 (8.5) | 63.0 (8.5) | 62.74 (8.49)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 7 | 13
  Male | 1093 | 1097 | 2190
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black | 93 | 77 | 170
  Hispanic | 52 | 71 | 123
  White | 926 | 931 | 1857
  Other | 27 | 25 | 52
  Unknown | 1 | 0 | 1
Urgent Status requiring surgery within 12 to 72 hours [Count of Participants; unit: Participants] | 146 | 146 | 292
Chronic obstructive pulmonary disease (COPD) [Count of Participants; unit: Participants] | 238 | 220 | 458
Peripheral vascular disease [Count of Participants; unit: Participants] | 163 | 179 | 342
Diabetes [Count of Participants; unit: Participants] | 491 | 470 | 961
Hypertension [Count of Participants; unit: Participants] | 952 | 948 | 1900
History of Depression [Count of Participants; unit: Participants] | 120 | 146 | 266

OUTCOME MEASURES:

1. Primary Outcome: Long-term All Cause Mortality Between On-pump and Off-pump Patients.
Description: Five-year mortality was initially assessed by matching the participants in the follow-up study to data in the VA Vital Status File and the National Death Index, which provided cause-of-death codes according to the International Classification of Diseases, 10th Revision.
Time Frame: 5 Years
Measure: Count of Participants; unit: Participants
Arm/Group | On-Pump | Off-Pump
Number analyzed (Participants) | 1099 | 1104
Participants
  All cause death | 131 | 168
  Composite MACE outcome with death | 298 | 342
  No MACE outcome | 670 | 594

2. Secondary Outcome: Long-term Major Adverse Cardiovascular Event (MACE) Between On-pump and Off-pump Patients
Description: Secondary outcomes included the 5-year rates of death from cardiac causes, repeat revascularization and nonfatal myocardial infarction.
Time Frame: 5 years
Measure: Count of Participants; unit: Participants
Arm/Group | On-Pump | Off-Pump
Number analyzed (Participants) | 1099 | 1104
Participants
  Death from cardiac causes | 58 | 70
  Acute myocardial infarction | 105 | 134
  Repeat revascularization procedure | 131 | 145
  Percutaneous coronary intrevention | 127 | 131
  Repeat Coronary artery bypass grafting (CABG) | 5 | 16
  No MACE outcome (non cardiac deaths included) | 673 | 608

ADVERSE EVENTS:
Time Frame: 5 Years
Arm/Group | On-Pump | Off-Pump
All-Cause Mortality (participants affected / at risk) | 131/1099 | 168/1104
Serious Adverse Events (participants affected / at risk) | 426/1099 | 496/1104
Other Adverse Events (participants affected / at risk) | 0/1099 | 0/1104
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | On-Pump (N=1099) | Off-Pump (N=1104)
Death from cardiac causes (Cardiac disorders) | 58 (58) | 70 (70)
Acute myocardial infarction (Cardiac disorders) | 105 (105) | 134 (134)
Repeat revascularization procedure (Cardiac disorders) | 131 (131) | 145 (145)
Percutaneous coronary intervention (Cardiac disorders) | 127 (127) | 131 (131)
Repeat Coronary artery bypass grafting (CABG) (Cardiac disorders) | 5 (5) | 16 (16)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes